CLINICAL TRIAL: NCT05795205
Title: Impact of Exercise on Metabolic Health Following Delayed Dinner Consumption in Healthy Adults
Brief Title: Delayed Dinner, Exercise and Glucose Metabolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan Normal University (Other)
Responsible Party: Principal Investigator, Yung-Chih Chen, Principal Investigator, National Taiwan Normal University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 202203HM008
Record Dates: First submitted 2023-03-21; First posted 2023-04-03 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Normal Dinner; Delayed Dinner; Exercise Plus Delayed Dinner
Keywords: late dinner; postprandial Glycaemia
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal dinner consumption (Experimental): Participants will have their dinner between 1800-1830pm
  Interventions: Behavioral: Normal dinner
- Delayed dinner consumption (Experimental): Participants will have their dinner between 2200-2230pm
  Interventions: Behavioral: Delayed dinner consumption
- Exercise with delayed dinner consumption (Experimental): Participants will exercise on a treadmill for 45 min followed by delayed dinner between 2200-2230pm
  Interventions: Behavioral: Exercise with delayed dinner consumption

INTERVENTIONS:
Behavioral: Normal dinner — Participants will consume breakfast at 0830-0855 am, lunch at 1230-1255 pm, followed by dinner at 1800-1825 pm. Snacks will be consumed at 2130-2140 pm.
  Arms: Normal dinner consumption
Behavioral: Delayed dinner consumption — Participants will consume breakfast at 08:30-08:55 am, lunch at 12:30-12:55 pm, followed by snacks at 18:00-18:10 pm. Dinner will be consumed at 21:30-21:55 pm.
  Arms: Delayed dinner consumption
Behavioral: Exercise with delayed dinner consumption — Participants will consume breakfast at 08:30-08:55 am, lunch at 12:30-12:55 pm, followed by snacks at 18:00-18:10 pm. Participants will exercise for 45 min at moderate-intensity 45 min prior to the delayed dinner at 21:30-21:55 pm.
  Arms: Exercise with delayed dinner consumption

SUMMARY:
This study aims to investigate whether exercise can alleviate the impact of delayed dinner on metabolic health next morning in sedentary healthy adults

ELIGIBILITY:
Inclusion Criteria:

* Physical inactive males
* Weight stable for more than 3 months (no change in weight +/- 3%)
* Non-smoker
* Able to walk comfortably on a treadmill
* Dinner consumers with normal sleep pattern (cycles)

Exclusion Criteria:

* Personal history of/existing diabetes, cardiovascular disease, metabolic disease or dyslipidaemia
* Taking medications that may influence lipid or carbohydrate metabolism or immune system function
* Unable to take part in exercise for any reason (e.g., injury or disability) or a positive response to any questions on the Physical Activity Readiness questionnaire (PAR-Q)

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 12 (Estimated)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-08-15 (Estimated); Study Completion 2023-08-15 (Estimated)

PRIMARY OUTCOMES:
Metabolic health (Oral glucose tolerance test, OGTT) | 120 minutes
  Fasting and postprandial blood glucose responses on next morning between trials
Metabolic health (Oral glucose tolerance test, OGTT) | 120 minutes
  Fasting and postprandial blood insulin responses on next morning between trials

SECONDARY OUTCOMES:
Inflammation | Baseline
  Fasting inflammatory biomarkers (IL-6, TNF-a, CRP) on next morning between trials
Visual analogue scale (VSA) | 120 minutes
  Changes in VAS from 0-100 mm (e.g., appetite & mood, etc.) on next morning between trials
Substate oxidation | 120 minutes
  Lipid and carbohydrate oxidation during OGTT between trials
Blood pressure | 120 minutes
  Changes in blood pressure (systolic and diastolic blood pressure) on next morning between trials
Appetite (lunch intake) | 30 minutes
  Ab libitum energy intake on next morning by the end of trial
HRV | Baseline
  Heart rate variability on next morning between trial
Gut hormones | 120 minutes
  Changes in blood gut hormones responses on next morning (e.g., GLP-1, PYY and GIP) between trials

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan Normal University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No